CLINICAL TRIAL: NCT03920514
Title: Different Timing of Intrauterine Insemination and Pregnancy Outcome in Patient With Unexplained Infertility :A Randomized Controlled Study
Brief Title: Timing and Intrauterine Insemination in Unexplained Infertility
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Salwa Sabry Ahmed Mohamed, Faculty of medicine sohag university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Intrauterine insemination
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Intrauterine Insemination
Keywords: infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Intervention Model Description: Women will be randomly divided in to four groups the first Group will undergo IUI after 24 H of hCG administration the second g will undergo IUI after 36 h after hCG the third Group will undergo IUI after 48h of hCG administration the last Group will undergo IUI at the time of hCG adminstration
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP 1 (Active Comparator): IUI 24 hours after hCGadminstration
  Interventions: Drug: hCG
- GROUP 2 (Active Comparator): IUI 36 hours after hCG adminstration
  Interventions: Drug: hCG
- GROUP 3 (Active Comparator): IUI 48 hours after hCG adminstration
  Interventions: Drug: hCG
- GROUP 4 (Active Comparator): IUI at time of hCG adminstration
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG — Women will be given hCG before or with IUI
  Other Names: Pregnyl

SUMMARY:
to determine the most suitable time for administration of (human chorionic gonadotropin )hCG prior to intrauterine insemination (IUI) to optimize pregnancy outcome and to have the best success rates so the cases divided in to four groups according to the time of hCG administration .

DETAILED DESCRIPTION:
IUI with or without ovarian stimulation is a common treatment for infertility ,it is a simple procedure the semen is prepared in the laboratory and transferred by a catheter and injected intrauterine .ultrasound folliculometry is used for monitoring follicular growth where some clinicians prefer the natural cycles and others prefer ovarian stimulation and human chorionic gonadotropin (hCG)trigger for better timing .so cases will take induction and folliculometry will be done until the follicle reach 18mm trigger with hCG .women will be randomly divided to four groups .the first group will undergo IUI at 24 after trigger the second IUI at36 hour after trigger the thirdG at 48 after trigger and finaly the last group IUI will be done simultaneos with trigger the out come the number of pregnant women for each group.

ELIGIBILITY:
Inclusion Criteria:

* Mild male infertility or unexplained infertility

Exclusion Criteria:

* Adanced male factor endometriosis uterine abnormality sever semen parameters i impairment according to WHO 2010 non ovulatory cycles bilatral tubal block

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 14 days after IUI
  Positive serum beta hCG test
Secondary outcome | 4 weeks after insemination
  Clinical pregnancy defined as prescence of at least one Intrauterine gestational sac with fetal pole on Transvaginal scan

CONTACTS AND LOCATIONS:
Overall Officials: Allam Mohamed Abd elmonam, Professor of obs and gyn, Principal Investigator — Faculty of medicine sohag university

REFERENCES:
- [Background] Aydin Y, Hassa H, Oge T, Tokgoz VY. A randomized study of simultaneous hCG administration with intrauterine insemination in stimulated cycles. Eur J Obstet Gynecol Reprod Biol. 2013 Oct;170(2):444-8. doi: 10.1016/j.ejogrb.2013.07.022. Epub 2013 Aug 6. PMID 23932307
- [Background] Cantineau AE, Janssen MJ, Cohlen BJ, Allersma T. Synchronised approach for intrauterine insemination in subfertile couples. Cochrane Database Syst Rev. 2014 Dec 21;2014(12):CD006942. doi: 10.1002/14651858.CD006942.pub3. PMID 25528596
- [Background] Yumusak OH, Kahyaoglu S, Pekcan MK, Isci E, Cinar M, Tasci Y. Does intrauterine insemination timing matter for achieving pregnancy during ovulation induction using gonadotropins? A retrospective cohort study. J Chin Med Assoc. 2017 Jun;80(6):366-370. doi: 10.1016/j.jcma.2016.06.005. Epub 2016 Sep 27. PMID 27686502